CLINICAL TRIAL: NCT01686074
Title: Motor Control in Chronic Fatigue Syndrome and Fibromyalgia.
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/679
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-02

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome
Keywords: Motor control; walking; physical activity; Muscle activity
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Chronic fatigue syndrome
- fibromyalgia
- chronic fatigue syndrome + fibromyalgia
- healthy sedentary control

SUMMARY:
This project is a comprehensive study, with main focus on motor control, comparing patients with chronic fatigue syndrome / myalgic encephalopathy (CFS/ME) and/or fibromyalgia syndrome (FMS). Focus of the present project will be on detailed movement analysis in a movement laboratory and involve functional tasks such as walking and standing. Investigations will also comprise muscle activity, reaction time and fine motor control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic fatigue syndrome or fibromyalgia

Exclusion Criteria:

* patients who already had been treated.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic fatigue syndrome and fibromyalgia from primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
motor control | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Egil A Fors, MD prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Avdeling for smerte og sammensatte symptomlidelser (ASSL) St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Rasouli O, Stensdotter AK, Van der Meer ALH. TauG-guidance of dynamic balance control during gait initiation in patients with chronic fatigue syndrome and fibromyalgia. Clin Biomech (Bristol). 2016 Aug;37:147-152. doi: 10.1016/j.clinbiomech.2016.07.008. Epub 2016 Jul 22. PMID 27474799
- [Result] Rasouli O, Fors EA, Borchgrevink PC, Ohberg F, Stensdotter AK. Gross and fine motor function in fibromyalgia and chronic fatigue syndrome. J Pain Res. 2017 Feb 7;10:303-309. doi: 10.2147/JPR.S127038. eCollection 2017. PMID 28223840